CLINICAL TRIAL: NCT03218878
Title: Pregnancy Outcomes Following Hysteroscopic Expansion of the Uterine Cavity for Patients With Small Cavities and Poor Reproductive Outcomes
Brief Title: Pregnancy Outcomes After Uterine Cavity Expansion
Status: Completed | Type: Observational
Sponsor: Reproductive Medicine Associates of New Jersey (Other)
Responsible Party: Sponsor
Other Study IDs: RMA-2017-04
Record Dates: First submitted 2017-07-13; First posted 2017-07-17 (Actual); Last update posted 2018-10-15 (Actual); Status verified 2018-10

CONDITIONS: Miscarriage; Uterus Abnormal; Infertility
MeSH Terms: conditions — Abortion, Spontaneous; Uterine Anomalies; Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study seeks to evaluate pregnancy outcomes following hysteroscopic uterine cavity expansion surgery for patients with dysmorphic uterine cavities and poor reproductive histories. Patients already planning to undergo surgery at the recommendation of their physicians will be recruited for participation.

DETAILED DESCRIPTION:
Any patient scheduled to undergo hysteroscopic expansion of the uterine cavity at RMANJ is eligible to participate in the study. Patients will be approached for consent to participate in the study prior to undergoing surgery. If enrolled, outcomes following surgery will be followed and recorded.

ELIGIBILITY:
Inclusion Criteria:

* Any patient scheduled to undergo hysteroscopic expansion of the uterine cavity

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients at an infertility clinic who are scheduled to undergo hysteroscopic expansion of the uterine cavity
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2017-07-21 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2018-09-10 (Actual)

PRIMARY OUTCOMES:
Ongoing pregnancy | 2 years
  presence of a fetal heartbeat at 8 weeks gestation

SECONDARY OUTCOMES:
Change in endometrial volume | 1 month
  Increase or decrease in endometrial volume post-operatively as assessed by saline sonography
Time to conceive | 2 years
  Time from post-operative visit to conception
Chemical pregnancy | 2 years
  Positive pregnancy test
Clinical pregnancy | 2 years
  Presence of a gestational sac on ultrasound
Pregnancy loss | 2 years
  Miscarriage; either biochemical or clinical pregnancy loss
Ectopic pregnancy | 2 years
  Pregnancy outside the uterus
Live birth | 2 years
  Delivery of a liveborn infant
Obstetrical complications | 2 years
  Any complications including hypertensive diseases, hemorrhage, etc.
Gestational age at delivery | 2 years
  in weeks and days
Birthweight | 2 years
  in grams

CONTACTS AND LOCATIONS:
Overall Officials: Linnea Goodman, MD, Principal Investigator — Reproductive Medicine Associates of New Jersey
Locations (1):
- Reproductive Medicine Associates of New Jersey, Basking Ridge, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Undecided